CLINICAL TRIAL: NCT03420963
Title: Ex-Vivo Expanded Allogeneic NK Cells for the Treatment of Solid Tumors of Pediatric Origin in Children and Young Adults
Brief Title: Donor Natural Killer Cells, Cyclophosphamide, and Etoposide in Treating Children and Young Adults With Relapsed or Refractory Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0085; NCI-2018-00909 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0085 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Cutaneous Melanoma; Recurrent Lip and Oral Cavity Carcinoma; Recurrent Malignant Endocrine Neoplasm; Recurrent Malignant Female Reproductive System Neoplasm; Recurrent Malignant Male Reproductive System Neoplasm; Recurrent Malignant Mesothelioma; Recurrent Malignant Neoplasm of Multiple Primary Sites; Recurrent Malignant Oral Neoplasm; Recurrent Malignant Pharyngeal Neoplasm; Recurrent Malignant Skin Neoplasm; Recurrent Malignant Soft Tissue Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Malignant Thyroid Gland Neoplasm; Recurrent Malignant Urinary System Neoplasm; Refractory Cutaneous Melanoma; Refractory Malignant Bone Neoplasm; Refractory Malignant Endocrine Neoplasm; Refractory Malignant Female Reproductive System Neoplasm; Refractory Malignant Male Reproductive System Neoplasm; Refractory Malignant Mesothelioma; Refractory Malignant Neoplasm of Multiple Primary Sites; Refractory Malignant Oral Neoplasm; Refractory Malignant Pharyngeal Neoplasm; Refractory Malignant Skin Neoplasm; Refractory Malignant Soft Tissue Neoplasm; Refractory Malignant Solid Neoplasm; Refractory Malignant Thyroid Gland Neoplasm; Refractory Malignant Urinary System Neoplasm
MeSH Terms: conditions — Melanoma; Mouth Neoplasms; Endocrine Gland Neoplasms; Mesothelioma, Malignant; Pharyngeal Neoplasms; Skin Neoplasms; Sarcoma; Thyroid Neoplasms; Urologic Neoplasms; Bone Neoplasms | interventions — Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, etoposide, NK cells) (Experimental): Patients receive cyclophosphamide IV QD over 30 minutes and etoposide IV QD over 60 minutes on days 1-5 in the absence of unacceptable toxicity. Patients then receive cord blood derived allogeneic NK cells IV on day 8.
  Interventions: Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells — Given IV
  Other Names: Allogeneic CB-derived Ex vivo-expanded NK Cells; CB-derived Expanded Allogeneic NK Cells; UCB-derived Expanded Allogeneic NK Cells; Umbilical Cord Blood-derived Expanded Allogeneic Natural Killer Cells
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16

SUMMARY:
This phase I trial studies the side effects and best dose of cord blood-derived expanded allogeneic natural killer cells (donor natural killer [NK] cells) and how well they work when given together with cyclophosphamide and etoposide in treating children and young adults with solid tumors that have come back (relapsed) or that do not respond to treatment (refractory). NK cells, white blood cells important to the immune system, are donated/collected from cord blood collected at birth from healthy babies and grown in the lab. Drugs used in chemotherapy, such as cyclophosphamide and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving NK cells together with cyclophosphamide and etoposide may work better in treating children and young adults with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety, maximum tolerated dose and/or recommended phase II dose of cord blood-derived expanded allogeneic natural killer cells (expanded allogeneic cord donor natural killer [NK] cells) following chemotherapy.

SECONDARY OBJECTIVES:

I. Determine the persistence of adoptively-transferred cord NK cells after solid tumor directed chemotherapy.

II. Preliminarily define the antitumor activity to adoptively transferred NK cells following the study preparative regimen in the confines of a phase I study.

III. Determine the immunophenotype and function of the infused NK cell product. IV. Preliminarily evaluate for any correlate of phenotype, killer cell immunoglobulin-like receptor (kir) haplotype, and function with overall response.

OUTLINE: This is a dose escalation study of cord blood derived allogeneic NK cells.

Patients receive cyclophosphamide intravenously (IV) once daily (QD) over 30 minutes and etoposide IV QD over 60 minutes on days 1-5 in the absence of unacceptable toxicity. Patients then receive cord blood derived allogeneic NK cells IV on day 8.

After completion of study treatment, patients are followed up at 3-4 days, and then every week for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* SCREENING: Patients with relapsed or refractory solid tumors and without known curative therapy or therapy proven to proven to prolong survival with acceptable quality of life.
* SCREENING: Patients older than 21 years must have a solid tumor considered by study doctor to be of the childhood cancer type.
* SCREENING: Performance level as measured by Karnofsky >= 60% for patients > 16 years of age or Lansky >= 60% for patients =< 16 years of age.
* SCREENING: Documentation of measurable or evaluable non-measurable disease.
* SCREENING: At least one documented histological verification of solid tumor diagnosis. Can be from original diagnosis or more recent.
* ENROLLMENT: Patient must have fully recovered (i.e. returned to baseline) from the clinically significant acute treatment-related toxicities of all prior treatments prior to beginning treatment on this protocol with exceptions of cytopenias resulting from persistent disease, hearing loss and alopecia.
* ENROLLMENT: Performance level as measured by Karnofsky >= 60% for patients > 16 years of age or Lansky >= 60% for patients =< 16 years of age.
* ENROLLMENT: Creatinine clearance >= 60 mL/min/1.73m^2 (calculated by 24 hour [h] urine collection or nuclear glomerular filtration rate [GFR] scan if 24 h collection is not possible) or a serum creatinine based on age and gender as follows:

  * Age, maximum serum creatinine (mg/dL):

    * 1 month to < 6 months, male 0.4, female 0.4;
    * 6 months to < 1 year, male 0.5, female 0.5;
    * 1 to < 2 years, male 0.6, female 0.6;
    * 2 to < 6 years, male 0.8, female 0.8;
    * 6 to < 10 years, male 1, female 1;
    * 10 to < 13 years, male 1.2, female 1.2;
    * 13 to < 16 years, male 1.5, female 1.4;
    * >= 16 years, male 1.7, female 1.4.
* ENROLLMENT: Adequate liver function, defined as: total bilirubin =< 2 mg/dl
* ENROLLMENT: Adequate liver function, as defined as serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x upper limit of normal (ULN) for age (unless Gilbert's disease or abnormal liver function due to primary disease).
* ENROLLMENT: Evidence of adequate bone marrow function (defined by absolute neutrophil count >= 750), unless patient has documented tumor metastasis to the bone marrow or other condition that results in cytopenia without abnormal marrow function.
* ENROLLMENT: Evidence of adequate bone marrow function (defined by platelets >= 50,000), unless patient has documented tumor metastasis to the bone marrow or other condition that results in cytopenia without abnormal marrow function.
* ENROLLMENT: Pulmonary symptoms controlled by medication and pulse oximetry >= 92% on room air.
* ENROLLMENT: Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the investigator. (Non-childbearing potential defined as pre-menarche, greater than one year post-menopausal or surgically sterilized).
* ENROLLMENT: Confirmation that a cord blood donor which is matched with the recipient at a 4, 5, or 6/6 human leukocyte antigen (HLA) class I (serological) and HLA class II (molecular) antigens.
* ENROLLMENT: Signed informed consent and if applicable pediatric assent.

Exclusion Criteria:

* SCREENING: Primary tumors of the central nervous system.
* SCREENING: Chronic corticosteroid dependence that is unable to be weaned to discontinue.
* SCREENING: Determined by study doctor that patient is unlikely to meet inclusion criteria after screening.
* ENROLLMENT: Uncontrolled arrhythmias or uncontrolled symptoms of cardiac disease noted by screening history and physical. Patients with known cardiac dysfunction should have an ejection fraction (EF) > 40% documented by echocardiogram (ECHO).
* ENROLLMENT: Patients where the burden of pulmonary metastasis, location, or bulkiness of disease may cause high morbidity if localized swelling such as causing uncontrolled symptoms, oxygen dependence, or location near a major bronchi as determined by investigator.
* ENROLLMENT: Pregnant females.
* ENROLLMENT: Any uncontrolled systemic infection.

Ages: 12 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the NK cell infusion
  Since toxicity is the primary outcome, patients with non-measurable disease (who are still evaluable) will be included in the analysis and in these cases standard methods for categorizing response of non-measurable disease will be used. Toxicity rate will be estimated separately by dose and cohort along with a 95% confidence interval. Adverse events will be tabulated for all the patients separately by dose levels.
Maximum tolerated dose and/or recommended phase 2 dose of cord blood-derived expanded allogeneic natural killer (NK) cells following chemotherapy | Up to 30 days after the NK cell infusion
  Primary analyses in this phase I trial are descriptive and exploratory. Toxicity rate will be estimated separately by dose and cohort along with a 95% confidence interval. Adverse events will be tabulated for all the patients separately by dose levels.

SECONDARY OUTCOMES:
Response rate per immune-related therapy trials Response Evaluation Criteria in Solid Tumors (irRECIST) | Up to 30 days after the NK cell infusion
  Complete response and partial response will be estimated separately by dose and cohort along with a 95% confidence interval. Correlation of NK cell persistence, phenotype, and function with overall response will be estimated using two-sample t-test/Wilcoxon sum-rank test and analysis of variance (ANOVA)/Kruskal-Wallis test as appropriate.
NK cell persistence, phenotype, and function | Up to 30 days after the NK cell infusion
  Correlation of NK cell persistence, phenotype, and function with overall response will be estimated using two-sample t-test/Wilcoxon sum-rank test and ANOVA/Kruskal-Wallis test as appropriate.
Overall survival (OS) | Up to 30 days after the NK cell infusion
  The Kaplan-Meier method will be used to estimate the distribution of OS. The description statistics of rate of OS may be analyzed separately by different tumor types and response/stable patients. Cox proportional hazards regression analysis may also be conducted to model the association between OS and factors of interest.
Time to progression (TTP) | Up to 30 days after the NK cell infusion
  The Kaplan-Meier method will be used to estimate the distribution of TTP. The description statistics of rate of TTP may be analyzed separately by different tumor types and response/stable patients. Cox proportional hazards regression analysis may also be conducted to model the association between TTP and factors of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios Petropoulos, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org